CLINICAL TRIAL: NCT06358105
Title: Simulator Training to Improve Interventional Cardiologist Skills (STARTERS) Trial
Acronym: STARTERS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Burzotta Francesco, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: id. 6457
Record Dates: First submitted 2024-04-02; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease
Keywords: simulation; training; fellows; coronary artery disease; coronary angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulator-based training group (Experimental): Interventional cardiology fellows will undergo a two-day training program on high-fidelity simulators
  Interventions: Procedure: Simulator-based training
- Standard group (Active Comparator): Interventional cardiology fellows will undergo standard training based on master-apprentice model
  Interventions: Procedure: Standard training

INTERVENTIONS:
Procedure: Simulator-based training — A two-day training program will be performed before starting their cath lab period as interventional cardiology fellows
  Arms: Simulator-based training group
Procedure: Standard training — Standard master-apprentice training interventional cardiology fellows' program during their cath lab period
  Arms: Standard group

SUMMARY:
The goal of this clinical trial is to learn if simulator-based training will improve interventional cardiology fellows' skills and will improve patient outcomes.

The main questions it aims to answer are:

* Does this training improve specific operative parameters recorded during initial coronary interventions performed as first operators under senior supervision?
* Will major and minor procedural complications be reduced after simulator-based training?

Interventional cardiology fellows in their first year of training will be randomized between standard master-apprentice training or simulator-based training before starting their cath lab period.

They will be supervised during their cath lab period as first operators by senior interventional cardiologists.

During their first 50 procedures performed as supervised first operator, specific procedural data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Specializing doctors who are about to start dedicated training in the interventional cardiology room
* Patients who must undergo coronary angiography examination.

Exclusion Criteria:

Specializing doctors:

* No interest in performing interventional cardiology procedures as first supervised operator (classical training)
* Experience as first supervised operator in interventional cardiology procedures
* Absence of informed consent

Patients:

* Acute Coronary Syndrome
* Severe left ventricular dysfunction with ejection fraction less than 30%
* Severe chronic renal failure (with glomerular filtration rate less than 30 ml/min)
* Absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Mean total fluoroscopy radiation time (expressed in seconds) | End of procedure
  Difference in Mean total fluoroscopy radiation time, during the periods where the cardiology fellows act as primary operators, between groups

SECONDARY OUTCOMES:
Mean arterial cannulation time (expressed in seconds) | End of procedure
  Difference in mean coronary cannulation time is considered as the time from sheath insertion to first right and left selective coronary angiography obtained (expressed in minutes)
Total radiation dose (expressed in cGy*cm2) | End of procedure
  Difference in total radiation dose adsorbed by patients as evaluated by dose-area product (DAP) (expressed in Gycm2)
Total contrast dose (expressed in ml) | End of procedure
  Difference in total contrast dose administered to the patients
Failure to achieve arterial cannulation (e.g.: rate of failure for each partecipant) | End of procedure
  Difference in failure to achieve arterial cannulation
Failure to achieve right coronary cannulation (e.g.: rate of failure for each partecipant) | End of procedure
  Difference in failure to achieve right coronary cannulation
Failure to achieve left coronary cannulation (e.g.: rate of failure for each partecipant) | End of procedure
  Difference in failure to achieve left coronary cannulation
Number of catheters used | End of procedure
  Difference in number of catheters used to complete the diagnostic procedure
Any major or minor procedural and clinical complication | Up to the end of index hospitalization or date of death from any cause (we collect any kind of clinical or procedural complication occuring during the determined period)
  Difference in any major or minor complication occurred during the procedure or the index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Burzotta, Prof, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Univrsitario Agostino Gemelli IRCCS, Rome, Italy

REFERENCES:
- [Background] Aggarwal S, Choudhury E, Ladha S, Kapoor PM, Kiran U. Simulation in cardiac catheterization laboratory: Need of the hour to improve the clinical skills. Ann Card Anaesth. 2016 Jul-Sep;19(3):521-6. doi: 10.4103/0971-9784.185548. PMID 27397459
- [Background] Pezel T, Coisne A, Bonnet G, Martins RP, Adjedj J, Biere L, Lattuca B, Turpeau S, Popovic B, Ivanes F, Lafitte S, Deharo JC, Bernard A. Simulation-based training in cardiology: State-of-the-art review from the French Commission of Simulation Teaching (Commission d'enseignement par simulation-COMSI) of the French Society of Cardiology. Arch Cardiovasc Dis. 2021 Jan;114(1):73-84. doi: 10.1016/j.acvd.2020.10.004. Epub 2021 Jan 5. PMID 33419690
- [Background] Sciahbasi A, Romagnoli E, Trani C, Burzotta F, Pendenza G, Tommasino A, Leone AM, Niccoli G, Porto I, Penco M, Lioy E. Evaluation of the "learning curve" for left and right radial approach during percutaneous coronary procedures. Am J Cardiol. 2011 Jul 15;108(2):185-8. doi: 10.1016/j.amjcard.2011.03.022. Epub 2011 Apr 29. PMID 21530937
- [Background] Joshi A, Wragg A. Simulator Training in Interventional Cardiology. Interv Cardiol. 2016 May;11(1):70-73. doi: 10.15420/icr.2016.11.1.70. PMID 29588710
- [Background] Popovic B, Pinelli S, Albuisson E, Metzdorf PA, Mourer B, Tran N, Camenzind E. The Simulation Training in Coronary Angiography and Its Impact on Real Life Conduct in the Catheterization Laboratory. Am J Cardiol. 2019 Apr 15;123(8):1208-1213. doi: 10.1016/j.amjcard.2019.01.032. Epub 2019 Jan 24. PMID 30732853
- [Background] Voelker W, Petri N, Tonissen C, Stork S, Birkemeyer R, Kaiser E, Oberhoff M. Does Simulation-Based Training Improve Procedural Skills of Beginners in Interventional Cardiology?--A Stratified Randomized Study. J Interv Cardiol. 2016 Feb;29(1):75-82. doi: 10.1111/joic.12257. Epub 2015 Dec 16. PMID 26671629